CLINICAL TRIAL: NCT03717376
Title: Specificity of Early Maladaptive Schemas in Functional Movement Disorders
Brief Title: Movement Disorders and Early Maladaptive Schemas
Acronym: SCHEMAF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18039J
Record Dates: First submitted 2018-10-15; First posted 2018-10-24 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-02

CONDITIONS: Functional Movement Disorder; Parkinson Disease; Dystonic Disorders
Keywords: Functional Movement Disorder; Functional Neurological Disorder; Early Maladaptive Scheme; Parkinson; Dystonia
MeSH Terms: conditions — Conversion Disorder; Parkinson Disease; Dystonic Disorders; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-questionnaire YSQ-S3 (Young Schema Questionnaire) — All participants will fill the YSQ-S3 at home and send it back to the main investigator.

SUMMARY:
Functional neurological disorders (FND) are neurological symptoms that cannot be explained by a lesion or related to an identified dysfunction of the central nervous system. FND are under-diagnosed, although common and highly disabling. Childhood trauma events are found in 30% to 80% of FND patients, and are more common in people with functional neurological disorder than in healthy controls and patient controls. Overall, risks factors, perpetuating factors and maintaining factors have been described in FND, although none of the studies have analysed the prevalence of Early Maladaptive Schemas (EMS) in these patients. EMS, as measured with the Young Schema Questionnaire (YSQ), are proposed to underlie a variety of mental health problems, in particular Personality Disorders. We hypothesize that some of these early maladaptive schemas may participate in the psychopathology and severity of FND.

The main outcome of this study is to assess the prevalence of early maladaptive schemas in patients presenting with Functional Movement Disorders in comparison to patients presenting with Parkinson's Disease or Organic Dystonia. The secondary outcomes are to further analyse the underlying relation of these early maladaptive schemas and (i) the severity of the motor symptoms, (ii) anxiety and/or depression, (iii) the occurrence of childhood trauma events in our participants.

DETAILED DESCRIPTION:
Functional neurological disorders (FND) are neurological symptoms that cannot be explained by a lesion or related to an identified dysfunction of the central nervous system. FND are under-diagnosed, although common and highly disabling. Functional Movement Disorders are a sub-category of FND, affecting the voluntary motor command. Childhood trauma events are found in 30% to 80% of FND patients, and are more common in people with functional neurological disorder than in healthy controls and patient controls. Overall, risks factors, perpetuating factors and maintaining factors have been described in FND, and some team research as Brown R. and al. have attempted to include it in psychopathological models such as the Integrative Conceptual Model in 2004. Nonetheless, none of the studies have analysed the prevalence of Early Maladaptive Schemas (EMS) in these patients. EMS, as measured with the Young Schema Questionnaire (YSQ), are proposed to underlie a variety of mental health problems, in particular Personality Disorders. Jeffrey Young has developed this concept in the 90's, through the so called "Schema Therapy". EMS are proposed as the core and main target for treatment of personality disorders and long-standing characterological problems. The current definition of an EMS is "a broad, pervasive theme or pattern, comprised of memories, emotions, cognitions, and bodily sensations, regarding oneself and one's relationships with others, developed during childhood or adolescence, elaborated throughout one's lifetime and dysfunctional to a significant degree". It has been studied in various conditions such as obesity, personality disorders, post-traumatic stress disorder, or obsessive-compulsive disorder, finding some EMS specificity in patients presenting with these conditions. In our study, we hypothesize that some of these early maladaptive schemas may participate in the psychopathology and severity of FND.

The main outcome of this study is to assess the prevalence of early maladaptive schemas in patients presenting with Functional Movement Disorders in comparison to patients presenting with Parkinson's Disease or Organic Dystonia. The secondary outcomes are to further analyse the underlying relation of these early maladaptive schemas and (i) the severity of the motor symptoms, (ii) anxiety and/or depression, (iii) the occurrence of childhood trauma events in our participants.

In order to reach these objectives, we aim to include 77 patients from which 30 patients with Functional Movement Disorder, 28 patients with Parkinson's disease, 19 patients with organic dystonia.

All eligible participants who have accepted to participate in the study will fill the YSQ-S3 (Short Form, French Version, validated and reliable instrument in clinical and research settings).The YSQ-S3 is a self-questionnaire which uses a Likert-type ranking, whereby 1 means "completely untrue of me" and 6 means "describes me perfectly". Similarly, questions range from life experiences to present feelings about certain situations. It consists of 90 self-report items, measuring all of the 18 EMS, aiming to describe one's functioning schemas over the past year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years-old
2. Being diagnosed with Parkinson's Disease (United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria) or with Functional Movement Disorder (Gupta & Lang criteria) or with Dystonia (criteria from Obeso et al. Mov Dis 2013)
3. Being previously included in the research protocol untitled " Retentissement des mouvements anormaux "
4. Patient informed and having given their non-opposition
5. Written and oral comprehension of French

Exclusion Criteria:

1. Pregnancy
2. Guardianship or Tutelage measure
3. Psychosis
4. Other neurological disorder (i.e.: brain tumor, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed-up at Pitié-Salpêtrière hospital with functional movement disorder, parkinson's disease or distonic disorders.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of early maladaptive schemas in patients with Functional Movement Disorders versus patients with Parkinson's Disease or Dystonic Disorders | Through study completion, an average of 1 year
  Score ≥16 in each schema on the Young Schema Questionnaire-S3 (YSQ-S3) is considered as pathological

SECONDARY OUTCOMES:
Correlation between the YSQ-S3 scores and the severity of motor symptoms (score from the Unified Parkinson's Disease Rating Scale (UPDRS) part 3) | Through study completion, an average of 1 year
  Clinical Severity score on UPDRS part 3 ranges from 0 (none) to 108 (severe)
Correlation between the YSQ-S3 scores and anxiety/depression symptoms (screened with the Hospital Anxiety and Depression Scale (HADS) together with the Mini International Neuropsychiatric Interview (MINI)) | Through study completion, an average of 1 year
  Presence of anxiety if HADS-Anxiety ≥10; Presence of depression if HADS-Depression ≥10
Correlation between the YSQ-S3 scores and self-reported childhood traumatic events (assessed with the Composite International Diagnosis Interview (CIDI) questionnaire) | Through study completion, an average of 1 year
  Assessment of the different types of childhood trauma events

CONTACTS AND LOCATIONS:
Overall Officials: Richard LEVY, MD. PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- APHP - Pitié-Salpêtrière hospital, Paris, France